CLINICAL TRIAL: NCT06375616
Title: A Comparative Study of Safety and Efficacy of Nafamostat Mesylate and Unfractionated Heparin in Renal Replacement Therapy for Sepsis Associated Acute Kidney Injury: A Randomized Controlled Trial
Brief Title: Comparison of Nafamostat and Unfractionated Heparin in RRT for Sepsis Associated AKI
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Shen Lei (Other)
Responsible Party: Sponsor-Investigator, Shen Lei, Chief Physician, Huashan Hospital
Organization: Huashan Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KY2024-023
Record Dates: First submitted 2024-04-15; First posted 2024-04-19 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Sepsis
Keywords: renal replacement therapy; acute kidney injury; nafamostat mesylate
MeSH Terms: conditions — Sepsis; Acute Kidney Injury | interventions — nafamostat; Injections; Heparin

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nafamostat (Experimental): Patients in NM arm will receive nafamostat mesylate as as anticoagulation during renal replacement therapy.
  Interventions: Drug: Nafamostat Mesylate
- Heparin (Active Comparator): Patients in UFH arm will receive unfractionated heparin as as anticoagulation during renal replacement therapy.
  Interventions: Drug: Unfractionated Heparin

INTERVENTIONS:
Drug: Nafamostat Mesylate — During RRT, a priming dose of 20 mg of nafamostat mesylate (NM) is administered before initiation of the procedure. Upon starting the machine, there is no loading dose, but a maintenance infusion rate of 25 mg/h of NM is maintained. NM is discontinued in the last half hour before the end of the RRT session.
  Other Names: Nafamostat; Nafamostat Mesylate for Injection; NM
  Arms: Nafamostat
Drug: Unfractionated Heparin — During RRT, a priming dose of 50 mg of unfractionated heparin (UFH) is administered before initiation of the procedure. Upon starting the machine, a loading dose of 0.2 mg/kg of UFH is given, followed by a maintenance infusion rate of 0.1 mg/kg/h of UFH. The anticoagulant is discontinued in the last half hour before the end of the RRT session.
  Other Names: heparin; UFH
  Arms: Heparin

SUMMARY:
The goal of this clinical trial is to compare the safety and efficacy of nafamostat mesylate (NM) and unfractionated heparin (UFH) in the process of renal replacement therapy (RRT) for patients suffering from sepsis associated acute kidney injury (SA-AKI). The main questions it aims to answer are:

The impact of NM and UFH on platelet count in septic patients undergoing RRT treatment.

The satisfaction with anticoagulation of NM and UFH in septic patients undergoing RRT treatment.

The 28-day all-cause mortality rate of septic patients undergoing RRT treatment with NM and UFH.

Researchers will use NM or UFH as anticoagulation during RRT in SA-AKI patients, assessing effects on platelet count, anticoagulation satisfaction, and mortality.

Participants will receive NM or UFH as anticoagulation during RRT for a minimum of 7 days. Bleeding symptoms, platelet count and coagulation function will be monitored daily. Platelet changes during the 7-day treatment period and survival status at 28 days post-treatment will be recorded.

DETAILED DESCRIPTION:
1. Research Description:

   This study is a prospective, randomized, parallel-controlled, blinded endpoint clinical trial. It aims to compare the safety and efficacy of NM and UFH in the process of RRT for septic patients.
2. Sample Size Calculation:

   The study design is an equivalence study. Based on relevant literature, the degree of platelet decrease caused by NM is approximately 20.9% ± 5%, and the degree of platelet decrease associated with UFH is approximately 23.3% ± 5%. The study compares the difference between these two rates at a significance level of 0.05 and a power of 80%. Therefore, the calculated sample size is 70 participants per group, with a 10% dropout rate considered, resulting in a total sample size of 156 participants (78 participants per group).
3. Adverse Event Recording:

   The adverse events in this study primarily include unplanned discontinuation of RRT (due to vascular access failure, filter clotting, or unstable vital signs). We will rigorously document the occurrence of adverse events and provide appropriate management. For serious adverse events resulting from platelet decrease, the study may be terminated early if platelet count drops below 25 × 10^9/L, decreases by more than 50% from baseline, or if active bleeding (digestive tract, skin mucosa, urinary tract, airway, etc.) occurs.
4. Statistical Analysis:

The intention-to-treat (ITT) population is defined as the set of patients who received at least one intervention after randomization. ITT analysis is the primary analysis for this study. The primary endpoint will be analyzed using analysis of covariance (ANCOVA). Anticoagulation satisfaction will be assessed using the Cochran-Mantel-Haenszel (CMH) test. The 28-day all-cause mortality rate will be analyzed using survival analysis, with survival described by Kaplan-Meier curves and compared by log-rank test. Cox regression will be used to assess the impact of NM and UFH on survival after adjusting for other confounding factors. A two-sided p-value <0.05 will be considered statistically significant.

5.Data Management and Confidentiality

1. Data Entry: Data entry and modifications will be performed by the researchers. The data should originate from original records and/or laboratory reports and must be consistent with the original documents. Any observations or examination results in the study should be entered into the forms promptly, accurately, completely, clearly, and in a standardized and truthful manner.
2. Participant Information Confidentiality Plan: All information regarding study participants must be kept strictly confidential. Participation in the study and any personal data collected during the study are considered confidential. Participant information and study data will be identified by a study identity number (ID number) rather than by name. Identifying information will not be disclosed to members outside the research team unless authorized by the participant. All research team members are required to maintain confidentiality regarding participant identities. Participant records will be stored in locked file cabinets accessible only to authorized research personnel. Government regulatory agencies or ethics committees may review participant data at the study site as required by regulations. When study results are published, no personal information about study participants will be disclosed.
3. Research Data Confidentiality Plan: Research data is also considered confidential. All research team members are required to maintain the confidentiality of research data and may not disclose research data to individuals outside the study team without permission from the principal investigator. Research data may not be transferred to external entities without permission from the hospital. Transfer of research data involving human genetic resources to foreign or domestically funded entities requires approval from the National Human Genetic Resources Administration unless the publication of research results meets legal requirements under normal circumstances.

6. Quality Control and Quality Assurance in Clinical Research: The primary investigator will organize relevant training to ensure the study is conducted according to protocol and adheres to Good Clinical Practice (GCP) principles. The completion of study records and other reports will also follow GCP principles and the research protocol. All data and materials must be traceable, and to ensure the reliability of research data, all observations and findings should be verifiable. Quality control will be applied at each stage of the study to ensure the reliability of all data and the accuracy of research procedures. The principal investigator will ensure that researchers adhere to the protocol, confirm the accuracy of data, and ensure the completeness of records and reports. Informed consent will be obtained from all participants before the study begins. Any deviations from the protocol will be promptly reported to the ethics committee. Standard operating procedures (SOPs) will be developed by the research team, and quality control procedures will be implemented at each stage of the study and data processing to ensure the standardization and reliability of study implementation and data operation.

7. Ethics Related to the Study: The interventions in both the experimental and control groups of this study are currently used clinical measures that do not impose additional burdens or costs on the subjects and involve no additional risks. This study is conducted under the premise of compliance with relevant Chinese regulations such as the "Ethical Review Methods for Biomedical Research Involving Humans" and international ethical guidelines such as the Helsinki Declaration.

8. Recruitment Methods: Patients admitted to the ward will be assessed by the researchers. Those who meet the inclusion and exclusion criteria will be enrolled by the researchers and will simultaneously sign an informed consent form. If a patient is conscious and capable of autonomous decision-making, they will personally sign the informed consent form. If a patient is unconscious or incapable of autonomous decision-making, an authorized representative will sign the informed consent form on their behalf.

Patients or their authorized representatives will be fully informed of the purpose and significance of this study, and that the interventions in both the experimental and control groups are currently used clinical measures that do not impose additional burdens, costs, or risks on the participants. Patients or their representatives will have sufficient time to consider their decision, and they will participate in the study only if they or their representatives fully understand the contents of the informed consent and voluntarily agree to participate.

9. Follow-up and Medical Measures after Study Completion: After the study concludes, treatment for the primary disease of the participants will continue as necessary. Patients will either continue hospitalization or be discharged after 28 days, and they will no longer be included in the follow-up schedule. For patients who experience serious adverse events (SAE) or significant medical events, the follow-up period may be extended to 40 days to ensure appropriate medical measures are taken after the study concludes.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 14 years old, and ≤ 90 years old.
* Sepsis or septic shock.
* AKI (Acute Kidney Injury), with stage of 2-3.
* Received renal replacement therapy (RRT) for ≥ 24 hours.
* Survival time ≥ 48 hours.

Exclusion Criteria:

* Presence of bleeding tendency or active bleeding.
* Pre-existing chronic kidney disease or already undergoing routine hemodialysis.
* With liver failure, severe hematologic disorders, malignancies, or other significant underlying diseases
* Pre-using of anticoagulant or antiplatelet medications such as aspirin, clopidogrel, rivaroxaban, dabigatran, or ticagrelor
* Allergy to heparin or nafamostat mesylate.
* Survival time < 48 hours or RRT treatment time < 24 hours.
* Initial platelet count < 50 × 10^9/L.
* Participation in another clinical trial within the past 1 month.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Estimated)
Dates: Start 2024-04 (Estimated); Primary Completion 2027-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Platelet decline rate | 7 days after initiation of RRT treatment
  (baseline platelet count - day 7 platelet count)/baseline platelet count *100%

SECONDARY OUTCOMES:
Satisfaction of filter anticoagulation | 7 days after initiation of RRT treatment
  using numbers 0-3 to evaluating the filter anticoagulation level, expressing as the median of all machines. (Grade 0: No clotting observed in the dialyzer after hemodialysis. Grade 1: Minimal clotting observed in approximately one-third of the dialyzer. Grade 2: Approximately half of the dialyzer shows clotting. Grade 3: The dialyzer is completely filled with clots.)

OTHER OUTCOMES:
All-cause mortality at 28 days | 28 days after initiation of RRT treatment
  survival or death condition of patients at 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Lei Shen, MD, Principal Investigator — Huashan Hospital
Locations (1):
- Huashan Hospital, Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zarbock A, Nadim MK, Pickkers P, Gomez H, Bell S, Joannidis M, Kashani K, Koyner JL, Pannu N, Meersch M, Reis T, Rimmele T, Bagshaw SM, Bellomo R, Cantaluppi V, Deep A, De Rosa S, Perez-Fernandez X, Husain-Syed F, Kane-Gill SL, Kelly Y, Mehta RL, Murray PT, Ostermann M, Prowle J, Ricci Z, See EJ, Schneider A, Soranno DE, Tolwani A, Villa G, Ronco C, Forni LG. Sepsis-associated acute kidney injury: consensus report of the 28th Acute Disease Quality Initiative workgroup. Nat Rev Nephrol. 2023 Jun;19(6):401-417. doi: 10.1038/s41581-023-00683-3. Epub 2023 Feb 23. PMID 36823168
- [Background] Poston JT, Koyner JL. Sepsis associated acute kidney injury. BMJ. 2019 Jan 9;364:k4891. doi: 10.1136/bmj.k4891. PMID 30626586
- [Background] Ohtake Y, Hirasawa H, Sugai T, Oda S, Shiga H, Matsuda K, Kitamura N. Nafamostat mesylate as anticoagulant in continuous hemofiltration and continuous hemodiafiltration. Contrib Nephrol. 1991;93:215-7. doi: 10.1159/000420222. No abstract available. PMID 1666354
- [Background] Uchino S, Bellomo R, Morimatsu H, Morgera S, Schetz M, Tan I, Bouman C, Macedo E, Gibney N, Tolwani A, Oudemans-van Straaten H, Ronco C, Kellum JA. Continuous renal replacement therapy: a worldwide practice survey. The beginning and ending supportive therapy for the kidney (B.E.S.T. kidney) investigators. Intensive Care Med. 2007 Sep;33(9):1563-70. doi: 10.1007/s00134-007-0754-4. Epub 2007 Jun 27. PMID 17594074
- [Background] Maruyama Y, Yoshida H, Uchino S, Yokoyama K, Yamamoto H, Takinami M, Hosoya T. Nafamostat mesilate as an anticoagulant during continuous veno-venous hemodialysis: a three-year retrospective cohort study. Int J Artif Organs. 2011 Jul;34(7):571-6. doi: 10.5301/IJAO.2011.8535. PMID 21786254
- [Background] Makino S, Egi M, Kita H, Miyatake Y, Kubota K, Mizobuchi S. Comparison of nafamostat mesilate and unfractionated heparin as anticoagulants during continuous renal replacement therapy. Int J Artif Organs. 2016 Jan;39(1):16-21. doi: 10.5301/ijao.5000465. Epub 2016 Feb 9. PMID 26868216